CLINICAL TRIAL: NCT06163911
Title: In-depth ECG Analysis for the Extraction of Biomarkers of Cardiac Mechanical Dispersion
Acronym: AFICIONADO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Olivier HUTTIN, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI117
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Pathology
MeSH Terms: interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No myocardial contractility abnormalities
  Interventions: Device: ECG; Device: Echocardiography
- Myocardial contractility abnormalities
  Interventions: Device: ECG; Device: Echocardiography

INTERVENTIONS:
Device: ECG — Routine care 12-lead electrocardiogram
Device: Echocardiography — Routine care echocardiography

SUMMARY:
Left ventricular systolic dysfunction (LVSD) refers to impaired contraction of the left ventricle, and can lead to heart failure and death. Early identification of LVSD, which often remains asymptomatic for years, is therefore crucial to mitigate the associated risks through appropriate treatment. Echocardiographic screening of asymptomatic individuals is costly, requires access to experts, and the criteria for selecting potential high-risk individuals for screening remain unclear.

Unlike echocardiography, the electrocardiogram (ECG) is a relatively low-cost procedure, routinely available and requiring little technical training to set up the examination and collect data, making it an interesting tool for early detection of LVSD.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and has not objected to the use of this data;
* Age ≥ 50;
* Persons who have undergone an echocardiographic examination and a 12-lead ECG examination during consultations at the CHRU de Nancy;
* Persons with at least one cardiovascular risk (obesity, diabetes, hypertension, etc.).

Exclusion Criteria:

* People with a history of heart disease (ischemic, valvular);
* Patients with significant 12-lead ECG abnormalities (complete bundle branch block, sequelae of myocardial infarction, etc.);
* ECG tracings or echocardiograms that cannot be analyzed.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen in consultation at the Cardiology Department of the Nancy CHRU who performed an echocardiography and a 12-lead ECG.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
F1 score for classification of cardiac contractility abnormalities | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, CHRU de Nancy, France